CLINICAL TRIAL: NCT02623270
Title: A Comparison of Controlled Ventilation With the V60 Non-Invasive Ventilator vs. Traditional Mask Ventilation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kai Kuck, Director of Bioengineering, Dept. of Anesthesiology, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00080301
Record Dates: First submitted 2015-07-29; First posted 2015-12-07 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Respiratory Complications Due to Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Noninvasive Ventilation (Experimental): After induction of anesthesia, checking of ability to bag mask ventilating the patient, the manual bag ventilation will be replaced by a Noninvasive Ventilator, V60 (Philips)
  Interventions: Device: Noninvasive Ventilator, V60 (Philips); Device: Manual Bag

INTERVENTIONS:
Device: Noninvasive Ventilator, V60 (Philips) — The noninvasive ventilator will be set to deliver 10 breaths per minute with a pressure setting of 8 cm H2O during exhalation and 20 cm H2O during inspiration. The inspired oxygen fraction given by the ventilator will be set at the maximum level (100% oxygen).
Device: Manual Bag — Oxygen will flow through the standard breathing circuit with the fresh gas flow rate set at 10 L/min and the patient will be ventilated. The anesthesia provider will manually bag mask ventilate the patient until the anesthesiologist feels comfortable that the patient can be ventilated appropriately.

SUMMARY:
The purpose of this study is to determine whether an experienced anesthesia provider can adequately and/or easily mask ventilate an anesthetized patient with a commercial non-invasive ventilator device.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether an experienced anesthesia provider can adequately and/or easily mask ventilate an anesthetized patient with a commercial non-invasive ventilator device. The ventilator subject of this study is commonly used in the ICU and investigators aim to evaluate its usefulness in the OR. Investigators believe that the ventilator will ventilate with consistent breath rates, adequate tidal volumes and minimal airway pressures. The providers subjective scoring of ease or difficulty of ventilation with each device will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* adults between 18-74 years of age,
* ASA status I-III,
* presenting for elective surgery requiring general anesthesia at the University of Utah
* able and will to provide informed consent

Exclusion Criteria:

* oropharyngeal or facial pathology,
* risk of aspiration (defined by need for rapid sequence intubation, uncontrolled gastroesophageal reflux disease),
* known and/or documented difficulty placing an endotracheal tube in the past,
* limited neck extension or flexion,
* restrictive lung disease,
* personal or familial history of malignant hyperthermia
* known or predicted severe respiratory disease or compromise.
* Female subjects must have a negative urine pregnancy screen.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Average of the difference in Respiratory Rate between Manual and Mechanical Ventilation (1/min) | Assessment will be made during the procedure during 10 consecutive breaths (depending on the breath rate, for approximately 1 minute) after induction but before intubation.
  Difference in average respiratory rate between manual ventilation and mechanical noninvasive ventilation averaged per patient, then averaged across all studied patients. Unit: 1/min.
Average of the difference in ideal body weight indexed tidal volume between Manual and Mechanical Ventilation (mL/kg) | Assessment will be made during the procedure during 10 consecutive breaths (depending on the breath rate, for approximately 1 minute) after induction but before intubation
  Difference in average tidal volume per ideal body weight between manual ventilation and mechanical noninvasive ventilation, averaged per patient, then averaged across all studied patients. Unit: mL/kg
In-Patient Average Difference of Standard Deviation in Respiratory Rate between Manual and Mechanical Ventilation (1/min) | Assessment will be made during the procedure during 10 consecutive breaths (depending on the breath rate, for approximately 1 minute) after induction but before intubation
  Difference in standard deviation of respiratory rate between manual ventilation and mechanical noninvasive ventilation averaged per patient, then averaged across all studied patients. Unit: 1/min.
In-Patient Average Difference of Standard Deviation in ideal body weight indexed tidal volume between Manual and Mechanical Ventilation (mL/kg) | Assessment will be made during the procedure during 10 consecutive breaths (depending on the breath rate, for approximately 1 minute) after induction but before intubation
  Difference in standard deviation of tidal volume per ideal body weight between manual ventilation and mechanical noninvasive ventilation, averaged per patient, then averaged across all studied patients. Unit: mL/kg

SECONDARY OUTCOMES:
Difficulty or ease of ventilation as perceived by anesthesia provider | Assessment will be made within one hour after the surgery has been completed.
  NASA TLX Score after each patient

CONTACTS AND LOCATIONS:
Overall Officials: Kai Kuck, Ph.D., Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data.

REFERENCES:
- [Derived] Fogarty M, Orr JA, Sakata D, Brewer L, Johnson K, Fang JC, Kuck K. A comparison of ventilation with a non-invasive ventilator versus standard O2 with a nasal cannula for colonoscopy with moderate sedation using propofol. J Clin Monit Comput. 2020 Dec;34(6):1215-1221. doi: 10.1007/s10877-019-00426-5. Epub 2019 Nov 23. PMID 31760586